CLINICAL TRIAL: NCT06241989
Title: Motivational Interviewing Supported Health Education on Digital Game Addiction and Cyberbullying inAdolescents Impact on Behavior
Brief Title: Digital Game Addiction and Cyberbullying in Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Professor, Facultyof Nursing, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023 - 1035
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Level of Digital Game Addiction; Level of Cyberbullying
Keywords: digital game addiction; cyberbullying; adolescent; motivational interview; health education
MeSH Terms: conditions — Cyberbullying; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive health education supported by motivational interviewing.
  Interventions: Other: health education supported by motivational interviewing
- Control (No Intervention)

INTERVENTIONS:
Other: health education supported by motivational interviewing — The intervention group will receive health education supported by motivational interviewing consisting of 6 sessions. Within the scope of the intervention, the first two sessions will be health education and the last four sessions will be motivational interviewing.
  Arms: Intervention

SUMMARY:
With the widespread use of technology and internet, digital game addiction and cyberbullying behaviors have increased among adolescents. Effective interventions are needed to prevent these behaviors. The aim of the study is to determine the effect of health education supported by motivational interviewing on digital game addiction and cyberbullying behaviors in adolescents. The research will be conducted with a randomized controlled trial design. The intervention group will receive six sessions of motivational interviewing-supported health education. Within the scope of the intervention, the first two sessions will be health education and the last four sessions will be motivational interviewing. It is planned that each session will be 35 minutes and the sessions will be implemented one week apart.

ELIGIBILITY:
Inclusion Criteria:

* Continuing 9th grade education
* Volunteering to participate in the research
* Being given permission by their families to participate in the study

Exclusion Criteria:

* Having problems understanding and speaking Turkish
* Visual-hearing impairment
* Having a neuropsychiatric disease

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Digital Game Addiction Scale-7 | baseline
  The scale consists of a total of seven items and has a five-point Likert scale. The respondent is asked to choose one of the options "never= 1", "rarely= 2", "sometimes= 3", "often= 4", "always= 5". The lowest score that can be obtained from the scale is 7 and the highest score is 35. Two methods, monothetic and polythetic, are used to determine the gaming addiction status. In the monothetic method, if the individual who answers the questionnaire gives a score of 3 (sometimes) or more to all items, and in the polythetic method, if he/she gives a score of 3 (sometimes) or more to at least four of all items, he/she is characterized as a game addict.
Revised Cyberbullying Inventory-II | baseline
  Participants answer the 10 items presented in two parallel forms twice on a 4-point scale (1 = never, 2 = once, 3 = two or three times, 4 = more than three times) to evaluate the cyberbullying behaviors they have done and been exposed to. The lowest score that can be obtained from the inventory is 10 and the highest score is 40. If the participants in the study mark any of the 10 items in the "I did it" section of the inventory with a score of at least "2 points = once" or higher, they are classified as "Cyber Bully". If the participants mark "1 point = Never" for all 10 items in the "I did it" section of the inventory, they are classified as "Never Cyberbullied".
Digital Game Addiction Scale-7 | first week
  The scale consists of a total of seven items and has a five-point Likert scale. The respondent is asked to choose one of the options "never= 1", "rarely= 2", "sometimes= 3", "often= 4", "always= 5". The lowest score that can be obtained from the scale is 7 and the highest score is 35. Two methods, monothetic and polythetic, are used to determine the gaming addiction status. In the monothetic method, if the individual who answers the questionnaire gives a score of 3 (sometimes) or more to all items, and in the polythetic method, if he/she gives a score of 3 (sometimes) or more to at least four of all items, he/she is characterized as a game addict.
Revised Cyberbullying Inventory-II | first week
  Participants answer the 10 items presented in two parallel forms twice on a 4-point scale (1 = never, 2 = once, 3 = two or three times, 4 = more than three times) to evaluate the cyberbullying behaviors they have done and been exposed to. The lowest score that can be obtained from the inventory is 10 and the highest score is 40. If the participants in the study mark any of the 10 items in the "I did it" section of the inventory with a score of at least "2 points = once" or higher, they are classified as "Cyber Bully". If the participants mark "1 point = Never" for all 10 items in the "I did it" section of the inventory, they are classified as "Never Cyberbullied".
Digital Game Addiction Scale-7 | twelfth week
  The scale consists of a total of seven items and has a five-point Likert scale. The respondent is asked to choose one of the options "never= 1", "rarely= 2", "sometimes= 3", "often= 4", "always= 5". The lowest score that can be obtained from the scale is 7 and the highest score is 35. Two methods, monothetic and polythetic, are used to determine the gaming addiction status. In the monothetic method, if the individual who answers the questionnaire gives a score of 3 (sometimes) or more to all items, and in the polythetic method, if he/she gives a score of 3 (sometimes) or more to at least four of all items, he/she is characterized as a game addict.
Revised Cyberbullying Inventory-II | twelfth week
  Participants answer the 10 items presented in two parallel forms twice on a 4-point scale (1 = never, 2 = once, 3 = two or three times, 4 = more than three times) to evaluate the cyberbullying behaviors they have done and been exposed to. The lowest score that can be obtained from the inventory is 10 and the highest score is 40. If the participants in the study mark any of the 10 items in the "I did it" section of the inventory with a score of at least "2 points = once" or higher, they are classified as "Cyber Bully". If the participants mark "1 point = Never" for all 10 items in the "I did it" section of the inventory, they are classified as "Never Cyberbullied".

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Çankaya/Türkiye, Turkey (Türkiye)